CLINICAL TRIAL: NCT00251147
Title: Prospective Randomized Study Comparing Open Acromioplasty and Rotator Cuff Repair Versus Arthroscopic Acromioplasty and Mini-Open Rotator Cuff Repair.
Brief Title: A Randomized Clinical Trial Comparing Open to Mini-Open Rotator Cuff Repair for Full-Thickness Rotator Cuff Tears.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Workers' Compensation Board, Alberta (Other); Canadian Orthopaedic Foundation (Other)
Responsible Party: Denise Chan, Orthopaedic Research Coordinator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10368
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff; open; arthroscopic; mini-open; acromioplasty; quality of life; shoulder
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Repair (Active Comparator)
  Interventions: Procedure: Open acromioplasty with rotator cuff repair
- Mini-open Repair (Active Comparator)
  Interventions: Procedure: Arthroscopic acromioplasty with mini-open repair

INTERVENTIONS:
Procedure: Open acromioplasty with rotator cuff repair — A standard vertical incision was made over the anterolateral aspect of the acromion. The deltoid muscle was split and stripped off the anterior aspect of the acromion. The anterior and inferior aspect of the acromion was removed. The coracoacromial ligament was excised. Repair of the tear in the cuff tendon(s) was accomplished by suturing leading edge of the tear into the greater tuberosity of the humerus at or near the original site of insertion of the cuff to bone. Trans-osseous sutures, suture anchors and tendon to tendon suture repair techniques were employed for a secure repair with the arm at the side. The surgeon was allowed to use whatever method(s) to create a secure repair. The deltoid was securely reattached to the acromion with the deltoid fascia repaired down the split.
  Other Names: Open repair
  Arms: Open Repair
Procedure: Arthroscopic acromioplasty with mini-open repair — A standard arthroscopic gleno-humeral arthroscopy was performed followed by an arthroscopic acromioplasty. Three standard arthroscopic portals were used. The lateral portal was centered in line with the cuff tear, and incorporated into the mini-open incision. Initially, a partial bursectomy was performed to improve visualization. The inferior surface of the anterior acromion and the coracoacromial ligament were removed. Following the arthroscopic acromioplasty, a 3-4cm lateral incision was performed in the area of the lateral portal. The deltoid muscle was split longitudinally to expose the tear in the rotator cuff. The tear was repaired in a similar manner to the open repair with tendon to tendon sutures, trans-osseous sutures and with suture anchors.
  Other Names: Mini-open repair; Scope mini-open
  Arms: Mini-open Repair

SUMMARY:
This study compares standard open rotator cuff repair versus arthroscopic mini-open rotator cuff repair by measuring the disease-specific quality of life at 2 years in patients with full thickness rotator cuff tears.

Hypothesis: There is no difference in disease-specific quality of life outcome at two years between open versus arthroscopic mini-open repair for patients with full-thickness rotator cuff tears.

DETAILED DESCRIPTION:
Rotator cuff injury affects a diverse group of patients and leads to significant disability with respect to lost time from work and the inability to play sports, thereby affecting the individual's quality of life.

The standard treatment for full-thickness rotator cuff repair is with an open acromioplasty procedure. An alternative procedure for a full-thickness rotator cuff tear is with a combined procedure of arthroscopic acromioplasty and mini-open repair, which has the potential advantages of a preserved deltoid origin, lower perioperative morbidity, shorter hospital stays and less soft tissue dissection. The progression towards arthroscopic repair requires a comparison to the standard, open procedure for full-thickness rotator cuff tears, using validated outcomes in a randomized fashion.

This study is designed as a multi-centre randomized controlled trial with a priori sample size calculation of 28 patients per group. Patients presenting with unremitting pain, failed conservative treatment of at least 3 months, weakness of the rotator cuff and positive imaging indicating a full-thickness rotator cuff tear are eligible for the study. Previous surgery on the affected shoulder and massive rotator cuff tears are excluded. Patients are randomized using computer-generated block randomization, stratified by surgeon, to either open or mini-open rotator cuff repair.

Disease-specific quality of life is assessed using the validated Rotator Cuff Quality of Life Questionnaire, a self-administered, 34-item questionnaire designed specifically to assess patients before and after surgery. It utilizes a visual analog scale scored out of 100, with a higher score reflecting a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unremitting pain in the affected shoulder who have failed conservative treatment for at least 3 months
* Weakness of rotator cuff (MRC grades 4-, 4 or 4+)
* Positive diagnostic imaging on the affected shoulder indicating a full-thickness rotator cuff tear which may include arthrogram, ultrasound or MRI
* Age > 18 years
* English speaking

Exclusion Criteria:

* A massive rotator cuff tear as demonstrated by Grade 3 or less muscle strength on testing internal and external rotation of the affected shoulder
* Previous surgery to the affected shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 1999-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Rotator Cuff Quality of Life Questionnaire (RC-QOL) | Baseline, 3, 6, 12, 24 months

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Score | Baseline, 3, 6, 12, 24 months
Shoulder Rating Questionnaire | Baseline, 3, 6, 12, 24 months
Functional Shoulder Elevation Test | Baseline, 6, 12, 24 months
Range of motion | Baseline, 3, 6, 12, 24 months
Strength | Baseline, 3, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hollinshead, MD, FRCSC, Principal Investigator — University of Calgary Sport Medicine Centre; Nicholas Mohtadi, MD, FRCSC, Principal Investigator — University of Calgary Sport Medicine Centre
Locations (4):
- Canada (4):
  - University of Calgary Sport Medicine Centre, Calgary, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Fowler Kennedy Sport Medicine Centre, London, Ontario
  - Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario